CLINICAL TRIAL: NCT02703857
Title: Study of Repeated Cefoxitin Administration in Major Abdominal Surgery Using a Microdialysis Technique
Acronym: PROPHYLOXITINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROPHYLOXITINE
Record Dates: First submitted 2016-02-09; First posted 2016-03-09 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Antibiotic Prophylaxis Surgery
MeSH Terms: interventions — Cefoxitin

INTERVENTIONS:
Drug: cefoxitin — Parenteral administration of 2g of cefoxitin at least 30 minutes before incision and then every 2 hours until closing

SUMMARY:
The surgical site infection is one of the most important causes of postoperative morbidity. The appropriate antibiotic prophylaxis is one of the most effective ways to prevent surgical site infections. The recommendations of the French Society of Anesthesia Resuscitation on antibiotic prophylaxis in long surgeries are based on low documentation, including frequency and dosage of reinjection.

The main objective of the study is to describe the tissue and plasma pharmacokinetics of cefoxitin after repeated injections.

This is an open monocentric study (phase 4) including adults aged 18 to 80 years in need of major abdominal surgery whose foreseeable time exceeds 4 hours and justifying an antibiotic prophylaxis by cefoxitin.

They receive 2 g cefoxitin parenterally at least 30 minutes before the incision and then every 2 hours until closing.

The primary endpoints are:

* Total and plasma free concentrations of cefoxitin 0, 10, 30, 60, 90, 120 minutes after start of each infusion cefoxitin
* Tissue free concentrations of cefoxitin every 20 minutes after the start of the first infusion cefoxitin until skin closure
* Urinary concentrations of cefoxitin

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent major abdominal surgery whose forseeable time exceeds 4 hours and requires an antibiotic prophylaxis by cefoxitin

Exclusion Criteria:

* morbid obesity (BMI > 35 kg/m²)
* severe renal impairment (clearance creatinine < 30ml/min)
* beta lactam hypersensitivity
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-20

PRIMARY OUTCOMES:
Total and free plasma of cefoxitin after repeated injections | 48 hours
Free tissue concentration of cefoxitin every 20 minutes after the beginning of injections | 48 hours
Concentration of cefoxitin in urine after every injection | 48 hours

SECONDARY OUTCOMES:
Percentage of time when tissue concentration of cefoxitin is higher than the minimal inhibitory concentration of target organisms | 48 hours
Concentrations of antibiotic in peritoneal fluid | 48 hours
Clearance of distribution of cefoxitin | 48 hours
Clearance of elimination of cefoxitin | 48 hours
Cmax of Cefoxitin | 48 hours
Vd of distribution o cefoxitin | 48 hours
Area under the curve of plasma and tissue concentration of cefoxitin | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Poitiers, Poitiers, France

REFERENCES:
- [Derived] Boisson M, Torres BGS, Yani S, Couet W, Mimoz O, Dahyot-Fizelier C, Marchand S, Gregoire N. Reassessing the dosing of cefoxitin prophylaxis during major abdominal surgery: insights from microdialysis and population pharmacokinetic modelling. J Antimicrob Chemother. 2019 Jul 1;74(7):1975-1983. doi: 10.1093/jac/dkz139. PMID 31220258